CLINICAL TRIAL: NCT03669237
Title: A Randomized Study From Single Institutions on Postoperative Bowel Function Following Sphincter Preservation Surgery in Patients With Rectal Cancer by Different Reconstruction Methods
Brief Title: Postoperative Bowel Function After SPS by Different Reconstruction Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YE Yingjiang (Other)
Responsible Party: Sponsor-Investigator, YE Yingjiang, Director of GI surgery department, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Bas-1904
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Bowel; Functional Syndrome
Keywords: Bowel Function; Sphincter Preservation Surgery; Reconstruction Method
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- end-to-side anastomosis (Experimental): All surgeries during the study were performed by the same experienced surgical team and were performed following TME principles. End-to-side anastomosis was used to perform colorectal anastomosis after primary tumor resection.
  Interventions: Procedure: different reconstruction methods
- end-to-end anastomosis (No Intervention): All surgeries during the study were performed by the same experienced surgical team and were performed following TME principles. After resection of the primary tumor, end-to-end anastomosis was used for colorectal anastomosis.

INTERVENTIONS:
Procedure: different reconstruction methods — Different reconstruction methods should be performed after sphincter preservation surgery in two groups.The methods include end-to-end anastomosis or end-to-side anastomosis
  Arms: end-to-side anastomosis

SUMMARY:
Colorectal cancer is one of the most common malignant tumors in the world. Surgery is still the main treatment for rectal cancer. With the popularization of stapler technology and the application of preoperative neoadjuvant therapy, more and more patients with rectal cancer have treated sphincter preservation surgery for rectal cancer. postoperative observation found that some patients with rectal cancer anus-preserving surgery had different degrees of defecation dysfunction after surgery, such as incontinence, tightness, increased frequency of bowel movements, and constipation. These clinical symptoms have been classified as "Low anterior resection syndrome (LARS)" in recent years.Now there is no treatment for LARS.Meanwhile,J-pouch and side-to-end anastomosis can help the patients,but there is few trials can prove this.This trial means to prove weather side-to-end anastomosis can improve bowel of rectal patients afer surgery.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common malignant tumors in the world. There are more than 1.7 million new cases worldwide each year, accounting for 9.7% of all cancers. Among them, 840,000 deaths, accounting for 8.5% of all cancer deaths, mortality Second only to lung cancer, liver cancer and gastric cancer. China is a country with high incidence of colorectal cancer, and its morbidity and mortality are the fifth highest in malignant tumors. Rectal cancer is the most common type of colorectal cancer. The incidence of rectal cancer in China is 14.0/100,000, which is the 7th cancer incidence rate in China.

Surgery is still the main treatment for rectal cancer. With the popularization of stapler technology and the application of preoperative neoadjuvant therapy, more and more patients with rectal cancer have treated sphincter preservation surgery for rectal cancer. The proportion of permanent ostomy has dropped to 16.9% to 29% . With the popularity of TME principles worldwide, the standardized treatment of rectal cancer is becoming more and more stable, and the postoperative survival rate of patients is steadily increasing. However, postoperative observation found that some patients with rectal cancer anus-preserving surgery had different degrees of defecation dysfunction after surgery, such as incontinence, tightness, increased frequency of bowel movements, and constipation. These clinical symptoms have been classified as "Low anterior resection syndrome (LARS)" in recent years. The research on LARS is still in its infancy, and its pathogenesis, influencing factors, pathophysiology and other explorations are not deep enough. Behind the various symptoms of low anterior resection syndrome is a complex pathophysiological basis. The symptoms and severity are affected by many changes in intestinal anatomy, nerve injury, postoperative healing process, diet structure and psychological status. The risk factors associated with the onset of defecation dysfunction after rectal cancer anal sphincter preservation include radiotherapy, total mesorectal excision, and tumor location. The role of various risk factors in the pathogenesis of defecation dysfunction after rectal cancer anal sphincter preservation is still controversial. At present, the diagnosis, grading and treatment of LARS are still in the exploration stage, and there is still no effective treatment.

Since the 1980s, a variety of colon-rectal anastomosis methods have been used in clinical practice to improve the dysfunction of rectal cancer after anal sphincter preservation, including J-pouch anastomosis, Colon transverse anastomosis, and end-to-side anastomosis. Each of the above three methods has its advantages and disadvantages: J-type storage bag improves the postoperative bowel movement anastomosis effect, but the technique is complicated and has more anastomotic symptoms; the colon transverse of the colon has a wide application range but the effect of improving the defecation function is poor; It has the longest history, but the time to apply to functional protection is the shortest, and there are few studies. Huttner et al published a meta-analysis published in 2015 (including 1636 cases from 21 clinical trials reports. Compared with end-to-end anastomosis, J-pouch can reduce the frequency of defecation and antidiarrheal drugs after 1 year after surgery. Similar results have been achieved with end-to-side anastomosis and colonic angioplasty; a review published by Brown et al also suggests that J-pouch can reduce the frequency of defecation and urgency of bowel movements during early (0-8 months) and mid-term (8-18 Months) .The end-to-side anastomosis achieved similar effects in each stage of the J-pouch, so it can be inferred that the end-to-side anastomosis (relative to end-to-end anastomosis) can improve postoperative defecation function. A retrospective study of end-to-end anastomosis and end-to-end anastomosis published in China also found that end-to-side anastomosis can reduce bowel movements and improve postoperative defecation function at 6 months after surgery. However, there is still no prospective clinical trial comparing the end-to-side anastomosis and end-to-end anastomosis for postoperative intestinal function. The ideal anastomosis should meet the characteristics of exact effect, simple operation and low complications. The end-to-side anastomosis is one of the potential choices, but its validity and safety lack relevant research evidence and need further study.

ELIGIBILITY:
Inclusion Criteria:

* The rectal adenocarcinoma is proved by pathology before surgery
* The lower margin of the tumor is less than 12cm higher from the anal verge under no anesthesia measured
* The tumor can be excised discussed by MDT
* Anus preserving operation can be performed
* ECOG score ranges between 0 and 2
* The estimate life is supposed to be more than 12 months
* The informed consent should be signed

Exclusion Criteria:

* The patient can not follow the experimental scheme
* The case is an emergency
* The patient is in pregnant or breast-feeding
* TME surgery can not be performed
* One-stage anastomosis can not be performed
* The patient has a history of anus surgery or rectal surgery
* The patient has a history of left hemicolectomy
* The patient has a long history of bowel dysfunction，such as diarrhea or dysporia before surgery
* The patient has cognitive disorder or communication disorder
* The patient has repeat infection or other disorders poorly controlled
* The patient joins other clinical trail that may disturb the bowel function

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Postoperative bowel function of 1 year after surgery | 1 year after surgery
  Each patients will be interviewed by telephone and asked to answer a copy of LARS score questionnaire.
  Designed for LARS patients only, the LARS score is a total score questionnaire containing five single choice questions with a corresponding score for each option. Each of the five questions tested a single symptom of the bowel function, including incontinence for flatus(score value from 0 to 7), incontinence for liquid stool (score value from 0 to 3), frequency of bowel movement (score value from 0 to 5), clustering of stools (score value from 0 to 11) and urgency (score value from 0 to 16). According to the total score of each patient, the questionnaire can evaluate the defecation function of the subject, which is divided into three categories from best to worst: no LARS (0 to 20), miner LARS (21 to 29) and major LARS (30 to 42).

SECONDARY OUTCOMES:
Operation safety | Data will be assess during operation and at the last visit before check-off.
  surgery time, blood loss, quality of surgical specimen, etc. will be record to assess safety of each reconstruction method.
  The incidence of key post-operative complication like anastomosis leakage, post-operative bleeding, server bowel obstruction, intra-abdominal abscess and surgical site infection, etc. will be record.
Postoperative bowel function within the first year | from the first month to the 11th month
  Each patients will be interviewed by telephone and asked to answer a copy of LARS score questionnaire.
  Designed for LARS patients only, the LARS score is a total score questionnaire containing five single choice questions with a corresponding score for each option. Each of the five questions tested a single symptom of the bowel function, including incontinence for flatus(score value from 0 to 7), incontinence for liquid stool (score value from 0 to 3), frequency of bowel movement (score value from 0 to 5), clustering of stools (score value from 0 to 11) and urgency (score value from 0 to 16). According to the total score of each patient, the questionnaire can evaluate the defecation function of the subject, which is divided into three categories from best to worst: no LARS (0 to 20), miner LARS (21 to 29) and major LARS (30 to 42).
Postoperative bowel function of the long stable result | 16 months after the primary surgery
  Each patients will be interviewed by telephone and asked to answer a copy of LARS score questionnaire after one year of operation.

CONTACTS AND LOCATIONS:
Overall Officials: Yingjiang Ye, M.D. ＆ PhD., Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided